CLINICAL TRIAL: NCT05565261
Title: Evaluation of Bite Force, Quality of Life, and Patients' Satisfaction of Edentulous Patients Using Complete Dentures and Implant-Supported Overdentures: An in Vivo Study
Brief Title: Evaluation of Bite Force, Quality of Life, and Patients' Satisfaction
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Esra Nur Avukat, Principal Investigator, Eskisehir Osmangazi University
Other Study IDs: EAvukat
Record Dates: First submitted 2022-06-23; First posted 2022-10-04 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Edentulous Jaw; Patient Satisfaction
Keywords: bite force; complete denture; implant supported overdentures; patient satisfaction; quality of life
MeSH Terms: conditions — Jaw, Edentulous; Patient Satisfaction | interventions — Denture, Complete

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Complete Dentures: The group consists of patients using conventional complete dentures applied to edentulous patients.
  Interventions: Device: complete denture
- Group 2: Implant Supported Overdentures: The group consists of patients who use implant-supported overdentures after 2 dental implants have been surgically placed in edentulous patients and osseointegration has occurred.
  Interventions: Device: complete denture

INTERVENTIONS:
Device: complete denture — Bite force was measured with a bite force measuring device. Quality of life and patient satisfaction were evaluated with questionnaires.

SUMMARY:
Objectives: The purpose of this study is to evaluate bite force (BF), oral health-related quality of life (OHRQoL), and patient satisfaction in 2-implant-supported overdentures. In addition, the effects of clinical parameters such as age, gender, implant length, implant diameter, locator attachment height, attachment color, and interimplant distance were also evaluated.

Material and Methods: A total of 51 patients were included in the study. BFs were measured with a force meter in complete dentures and implant-supported overdentures. OHRQoL was assessed with the Oral Health Impact Profile (OHIP-14) and patient satisfaction was assessed with the Visual Analog Scale (VAS).

DETAILED DESCRIPTION:
New complete dentures with bilateral balanced occlusion were fabricated for the patients. The patients wore the prosthesis for at least 8 weeks to allow the muscles to adapt. After adaptation to the dentures, 2 dental implants (Astra Tech Implant System, Dentsply Sirona) were placed in the interforaminal region of the mandible. A minimum of 3 months was waited for the dental implants to osseointegrate. After osseointegration, a clinical examination of the prostheses was performed. The clinical examination evaluated the accuracy of the prostheses in terms of occlusion and vertical dimension, their adaptation to the tissue, and the health of the soft tissue. If cracks or fractures were present, the prosthesis was repaired, and if a defect in tissue adaptation was detected, the prostheses were idealized by relining. The OccluSense® computerized occlusion analysis system (Dr. Jean Bausch GmbH & Co. KG, Cologne, Germany) was used to check occlusion evaluation, masticatory force distribution, and premature contact due to wear. In the case of premature contact, contacts were eliminated and the first bite force (BF) values of patients with correct occlusion were measured. The maximum BF was measured with a forcemeter (Akson, Istanbul, Turkey). The intraoral sensor of the device was placed unilaterally at the level of the 1st molar. To ensure stability, a bite block of the same thickness was placed in the contralateral dental arch. Patients were seated in a comfortable position with the Frankfurt horizontal plane parallel to the horizontal plane. Patients were asked to bite hard for 3 seconds and the measurement was repeated 3 times. To obtain a reliable value, patients rested for 1 minute after each measurement. The maximum BF was accepted as the highest value among the three bite forces. The mean value of the unilateral right and left measurements was used for data analysis. After measurement, the dentures were attached to the Locator Attachments (Zest Anchors LLC, Escondido, USA). Patients had to wait at least 8 weeks to adapt to the implant-supported overdentures. After the adaptation period, the second BF values of the patients wearing complete dentures in the maxilla and implant-supported overdentures in the mandible were measured.

Oral health-related quality of life and patients satisfaction In this phase, patients were asked to complete the OHIP-14 questionnaires to assess their quality of life and VAS forms to assess patient satisfaction. To assess the impact of clinical parameters, age, gender, implant lengths, implant diameters, locator attachment height, attachment color, and interimplant distance were also recorded.

OHRQoL was assessed using the Turkish version of the Oral Health Impact Profile (OHIP-14). Patients were asked to indicate how often the corresponding OHIP parameter occurred in the past month. OHIP-14 contains 14 questions related to 7 different main topics. The 7 main themes are functional limitations, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Patients answered the questions as 0 = Never, 1 = Rarely, 2 = Occasionally, 3 = Quite often, and 4 = Frequently. Scoring was based on 7 main categories and 8 data as the sum of all these categories. The total score of the OHIP-14 is at least 0 and the highest score is 56. A low score at the end of the test indicates a positive impact on OHRQoL, while a high score indicates a negative impact.

Patient satisfaction was measured with the questionnaire VAS. The questions in the questionnaires evaluated the comfort of the prosthesis, convenience in chewing, aesthetics, speech, stability, and ease of cleaning. Patients answered the questions with 5=Totally satisfied, 4=Satisfied, 3=Adequate, 2=Not satisfied, 1=Not at all satisfied. Higher scores indicate higher patient satisfaction.

ELIGIBILITY:
Inclusion criteria:

* Patients without pathology in intraoral tissues
* Patients who have not experienced implant loss until the prosthesis stage
* Patients without any systemic disease that would endanger the prognosis of the implant
* Patients with good bilateral balanced occlusion
* Patients who could understand and answer the questions in the questionnaire were included in the study.

Exclusion Criteria:

* Patients with parafunctional habits
* Patients with masticatory muscles or temporomandibular joint complaints
* Patients using drugs that affect muscle activity
* Patients who did not come to the control session on time were excluded from the study.

Ages: 47 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who were completely edentulous were included in the study.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Bite force | December 2019-January 2022
  Bite force in Newton
Interimplant distance | December 2019-January 2022
  Interimplant distance in millimeters
The height of the locator attachment | December 2019-January 2022
  The height of the locator attachment is in millimeters.
Quality of Life | December 2019-January 2022
  Quality of Life was assessed using the Oral Health Impact Profile(OHIP-14) (0-4 units, 0 for never to 4 for always).
Patient satisfaction | December 2019-January 2022
  Patient satisfaction was assessed using the VAS(visual analogue scale, 1-5 units, 1 not satisfied to totally satisfied).
Dental implant length | December 2019-January 2022
  Dental implant length in millimeters
Dental implant diameter | December 2019-January 2022
  Dental implant diameter in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Esra Avukat, Principal Investigator — Research Assistant
Locations (1):
- Esra Nur Avukat, Odunpazari, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feine JS, Carlsson GE, Awad MA, Chehade A, Duncan WJ, Gizani S, Head T, Heydecke G, Lund JP, MacEntee M, Mericske-Stern R, Mojon P, Morais JA, Naert I, Payne AG, Penrod J, Stoker GT, Tawse-Smith A, Taylor TD, Thomason JM, Thomson WM, Wismeijer D. The McGill consensus statement on overdentures. Mandibular two-implant overdentures as first choice standard of care for edentulous patients. Gerodontology. 2002 Jul;19(1):3-4. No abstract available. PMID 12164236
- [Result] Thomason JM, Feine J, Exley C, Moynihan P, Muller F, Naert I, Ellis JS, Barclay C, Butterworth C, Scott B, Lynch C, Stewardson D, Smith P, Welfare R, Hyde P, McAndrew R, Fenlon M, Barclay S, Barker D. Mandibular two implant-supported overdentures as the first choice standard of care for edentulous patients--the York Consensus Statement. Br Dent J. 2009 Aug 22;207(4):185-6. doi: 10.1038/sj.bdj.2009.728. PMID 19696851
- [Result] Mumcu E, Bilhan H, Geckili O. The effect of attachment type and implant number on satisfaction and quality of life of mandibular implant-retained overdenture wearers. Gerodontology. 2012 Jun;29(2):e618-23. doi: 10.1111/j.1741-2358.2011.00531.x. Epub 2011 Jul 4. PMID 21726276
- [Result] Muller F, Duvernay E, Loup A, Vazquez L, Herrmann FR, Schimmel M. Implant-supported mandibular overdentures in very old adults: a randomized controlled trial. J Dent Res. 2013 Dec;92(12 Suppl):154S-60S. doi: 10.1177/0022034513509630. Epub 2013 Oct 24. PMID 24158342
- [Result] Wang Y, Baumer D, Ozga AK, Korner G, Baumer A. Patient satisfaction and oral health-related quality of life 10 years after implant placement. BMC Oral Health. 2021 Jan 14;21(1):30. doi: 10.1186/s12903-020-01381-3. PMID 33446161
- [Result] Enkling N, Saftig M, Worni A, Mericske-Stern R, Schimmel M. Chewing efficiency, bite force and oral health-related quality of life with narrow diameter implants - a prospective clinical study: results after one year. Clin Oral Implants Res. 2017 Apr;28(4):476-482. doi: 10.1111/clr.12822. Epub 2016 Mar 24. PMID 27009835